CLINICAL TRIAL: NCT06534723
Title: A 12-month Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Clinical Trial of Wujia Yizhi Granules in the Treatment of Mild-to-moderate Alzheimer's Dementia (Syndrome of Deficiency of Spleen and Kidney).
Brief Title: Phase 3 Clinical Trial of Wujia Yizhi Granules in the Treatment of Mild-to-moderate Alzheimer's Dementia (Syndrome of Deficiency of Spleen and Kidney)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Jishengtang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH110-60101
Record Dates: First submitted 2024-07-03; First posted 2024-08-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wujia Yizhi Granules (Experimental): Participants received Wujia Yizhi Granules 6g ,BID,once in the morning and once in the evening, at an interval of more than 8 hours, for up tp 12 months.
  Interventions: Drug: Wujia Yizhi granules
- Placebo (Placebo Comparator): Participants received Wujia Yizhi granules simulator 6g ,BID,once in the morning and once in the evening, at an interval of more than 8 hours, for up tp 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Wujia Yizhi granules — Drug: Wujia Yizhi granuless
  Arms: Wujia Yizhi Granules
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled phase 3 design aimed at further verifying the safety and efficacy of Wujia Yizhi granules for mild-to-moderate Alzheimer's dementia

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled phase 3 clinical trial targeting patients with mild-to-moderate Alzheimer's dementia (TCM differentiated as syndrome of deficiency of spleen and kidney). 570 subjects were recruited and randomly assigned to the experimental and placebo groups at a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age range : 50 - 80 years old.
2. Informed consent signed and dated by patient or legal representative.
3. The participants are mild-to-moderate AD patients who meet the diagnostic criteria for AD proposed by the National Institute on Aging and the Alzheimer's Association (NIA-AA) in 2018 and have a disease course of more than 6 months. If participants lack previous pathological evidence or biomarkers of Alzheimer's dementia, they must have evidence of β-amyloid deposition biomarkers during screening (PET with abnormal amyloid deposition or low cerebrospinal fluid Aβ 42 and Aβ 42/Aβ 40 ratio).
4. MMSE score 11 to 26;CDR-GS score 1 to 2 。

Exclusion Criteria:

1. Participants with non AD induced memory and cognitive impairment, such as diagnosis of other types of dementia, including but not limited to mixed dementia (AD VaD), vascular dementia (VD), Parkinson's disease dementia (PDD), Lewy body dementia (DLB), Huntington's disease related dementia, frontotemporal lobe dementia (FTD), etc; Endocrine system disorders (such as thyroid diseases, parathyroid diseases) and dementia caused by folate, vitamin B12 deficiency, or any other reason; Existence of consciousness disorders, etc.
2. Participants have a history of epileptic seizures.
3. Participants are psychiatric patients, including but not limited to schizophrenia, affective schizophrenic disorder, bipolar disorder, or delirium.
4. HAMD-17 score ≥ 17 points.
5. HAMA score ≥ 14 points.
6. Participants were taking antidepressants, anxieties, and antipsychotic drugs during screening.
7. HIS score ≥ 4 points..

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to endpoint in Alzheimer's dementia Assessment Scale-Cognitive subscore (ADAS-Cog12). | Change from Baseline to Month 12
  The Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS-Cog12) is used to assess the cognitive function level of AD subjects. The ADAS-Cog12 score range is 0-75 points, and the higher the score on the scale, the more severe the cognitive impairment.
Change from baseline to endpoint in Clinical Dementia Rating-Sum of Boxes (CDR-SB). | Change from Baseline to Month 12
  The Alzheimer's Disease Assessment Scale - Cognitive Scale (CDR-SB) is used to assess the cognitive function level of AD subjects. The CDR-SB score range is 0-3 points, and the higher the score on the scale, the more severe the cognitive impairment.

SECONDARY OUTCOMES:
Change from baseline to endpoint in ADAS-Cog12. | Change from Baseline to month 3, 6, and 9
  The Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS-Cog12) is used to assess the cognitive function level of AD subjects. The ADAS-Cog12 score range is 0-75 points, and the higher the score on the scale, the more severe the cognitive impairment.
Change from baseline to endpoint in CDR-SB. | Change from Baseline to month 3, 6, and 9
  The Alzheimer's Disease Assessment Scale - Cognitive Scale (CDR-SB) is used to assess the cognitive function level of AD subjects. The CDR-SB score range is 0-3 points, and the higher the score on the scale, the more severe the cognitive impairment.
Change from baseline to endpoint in he Alzheimer's dementia Cooperative Study-Activities of Daily Living (ADCS-ADL) scale. | Change from Baseline to month 3, 6, 9 and 12
  The Alzheimer's Disease Collaborative Study Group - Activities of Daily Living Scale (ADCS-ADL) is used to evaluate the daily living abilities of AD subjects. The score range of ADCS-ADL is from 0 to 78, with higher numbers indicating better daily functioning.
Change from baseline to endpoint in Mini-Mental State Examination (MMSE). | Change from Baseline to month 3, 6, 9 and 12
  The Simple Intelligent State Examination Scale (MMSE) has a total of 19 items, with scores ranging from 0 to 30. In clinical practice, the diagnostic threshold is usually adjusted based on educational level, with university ≤ 26 points, middle school ≤ 24 points, primary school ≤ 23 points, and illiteracy ≤ 22 points, indicating dementia.
Change from baseline to endpoint in Neuropsychiatric Inventory (NPI). | Change from Baseline to month 3, 6, 9 and 12
  The Neuropsychiatric Inventory (NPI) includes a total of 12 items in 10 behavioral domains and 2 autonomic nervous system domains, with a score range of 0-144. The caregiver distress rating is 0-60, where 0 represents the best, and the higher the score, the higher the level of distress.
Change from baseline to endpoint in Traditional Chinese Medicine Syndrome Score | Change from Baseline to month 3, 6, 9 and 12
  TCM syndrome scale was used to evaluate the changes of TCM symptoms and signs before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Chen, Medical Doctor, Principal Investigator — Fujian Medical University Affiliated Union Hospital
Locations (1):
- Fujian Medical University Affiliated Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No